CLINICAL TRIAL: NCT06819189
Title: Role of Metal Ion Transporter ZIP8 in Alcohol Related Behaviors
Brief Title: Role of Metal Ion Transporter ZIP8 in Alcohol-Related Behaviors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10002228; 002228-AA
Record Dates: First submitted 2025-02-08; First posted 2025-02-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01-08

CONDITIONS: Healthy Volunteer
Keywords: Alcohol
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IV Ethanol (Other): IV Ethanol
  Interventions: Drug: Ethanol

INTERVENTIONS:
Drug: Ethanol — IV Ethanol

SUMMARY:
Background:

Alcohol use disorder (AUD) can damage people s health, work, and family. Researchers want to know more about why some people are more vulnerable to AUD than others. The ZIP8 gene may be linked to an increased risk of AUD. Researchers want to find out how different forms of the ZIP8 gene affect how healthy people drink alcohol and how alcohol affects their brain.

Objective:

To study how genes may affect how people drink alcohol and how it affects their brain.

Eligibility:

Healthy people aged 21 to 60 years. They must not smoke, and they must have no history of AUD. They must have European ancestry and be enrolled in Natural History Protocol (14-AA-0181).

Design:

Participants will have 2 study visits.

At the first visit, participants will be given alcohol; it will be infused through a tube attached to a needle inserted into a vein. They may self-administer each dose by pressing a button. Over time, they will have to press the button an increasing number of times to receive more alcohol. The infusion period will last 2.5 hours.

Participants will have blood samples taken and breath measurments, and they will do computer tasks and complete questionnaires during and after the infusion. After the infusion, they will remain in the clinic until their breath alcohol levels drop to a safe level.

At the second visit, participants will have an imaging scan of their brain. They will do tasks and play games on a computer screen during the scan.

Some participants may have an extra visit for screening. A mid-study visit may also be needed if more than 6 months pass between the 2 study visits....

DETAILED DESCRIPTION:
Study Description:

Genome-wide association studies of alcohol use disorder and alcohol consumption phenotypes have consistently identified significant associations with the metal ion transporter ZIP8 gene, specifically a single nucleotide polymorphism SLC39A8. The goal of this study is to examine the effect of SLC39A8 variation on alcohol-related phenotypes using an integrated translational pharmacogenetics approach. Alcohol-seeking and consumption will be evaluated using a human lab model of alcohol self-administration in a sample of 50 male and female non-AUD drinkers, classified into 2 groups based on their SLC39A8 genotype (rs13107325): 1) T-allele carriers (TT or CT genotype), and 2) CC-allele homozygotes (CC genotype). Participants will also undergo resting-state functional MRI scanning to assess functional connectivity in brain networks such as the salience network, and task-based functional MRI scans to assess activation in brain regions associated with reward processing and decision making, for association with SLC39A8 SNP genotype. The hypotheses guiding this project are that SLC39A8 variation would be associated with altered alcohol self-administration phenotypes of alcohol seeking and consumption, as well as with brain activation in brain regions associated with reward and decision making that are also associated with alcohol s effects.

Objectives:

Primary Objective:

To examine the effect of SLC39A8 genetic variation on IV alcohol self-administration phenotypes in non-AUD drinkers.

Secondary Objective:

To examine the effect of SLC39A8 genetic variation on brain activation and responses using functional magnetic resonance imaging in non-AUD drinkers.

Endpoints:

Primary Endpoints:

IV alcohol self-administration measures - Peak breath alcohol concentration (BrAC), number of alcohol infusions received.

Secondary endpoints:

brain activation (fMRI BOLD signal change) associated with reward during the monetary incentive delay (MID) task. Brain activation (fMRI BOLD signal change) associated with decision making during the risk task. Brain regions of interest include striatum, insula, cingulate cortex and prefrontal cortex.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male and female participants between 21-60 years of age. [Based on: identification provided to Clinical Center Admissions office].
  2. Non-smokers with no history of smoking in the past year and not a daily smoker for more than 1 month in their lifetime. [Based on: smoking history questionnaire, Additional History Form]
  3. Participants of European ancestry: the minor T allele of rs13107325, has a frequency of 0.08 in European ancestry, but is almost absent in Asian and African populations (http://www.ensembl.org). Due to the rare occurrence of the T allele and to avoid populations stratification in this small sample-sized study, only participants with self-reported White racial category (European ancestry) will be enrolled in this study.
  4. Inclusion criteria for persons of childbearing potential: Use of adequate method of birth control during the study, if participant is sexually active and is not surgically sterilized. Adequate methods of contraception include use of oral contraceptives; use of barrier method of contraceptive; use of an approved IUD or other long-acting reversible contraceptive (LARC); have a male sexual partner who is surgically sterilized; or have exclusively same-sex sexual partner(s). Justification: To minimize the risk of administering alcohol to pregnant persons of childbearing potential, given the known effects of alcohol exposure on fetuses. [Based on: medical history].
  5. Ability to understand the written consent form and willing to sign it. [Based on: consent quiz].

EXCLUSION CRITERIA:

1. Current history (past 12 months) of major medical illness, including CNS, cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders, or positive hepatitis (A, B antigen, or C), or HIV test. Justification: Many illnesses may alter the neuropsychological effects of alcohol as well as MRI measures. Hepatitis can alter liver function and alcohol pharmacokinetics. HIV infection can alter brain function. [Based on: clinically significant findings on medical history and physical exam, ECG, laboratory tests].
2. Current history of psychiatric disorders, including depressive disorder, bipolar disorder, or anxiety disorders. Justification: Concurrent psychopathology can alter brain function and alcohol response. [Based on: SCID interview]
3. Lifetime history of psychotic disorders, obsessive compulsive disorder (OCD), posttraumatic stress disorder (PTSD), or eating disorder. Justification: These disorders can have long-term effects on brain function and alcohol response. [Based on: SCID interview]
4. Current or lifetime diagnosis of alcohol or substance use disorder. Past mild AUD or past mild SUD with no current symptoms for at least 2 years will not be exclusionary. Justification: History of moderate to severe alcohol or substance use disorder will impact brain function and alcohol response We do not anticipate past mild AUD or SUD in remission for 2+ years would have such impact on brain function and alcohol response. We will examine this in an exploratory analysis. We will also do a follow-up telephone/telehealth visit with these participants to assess any changes in alcohol or substance use or problems related to their participation in the study. [Based on: SCID interview].
5. Currently seeking treatment for alcohol use disorders. Justification: It would be unethical to administer alcohol to individuals seeking treatment for alcohol problems. Also, this study does not provide treatment for individuals with alcohol use disorder. [Based on: medical history]
6. Non-drinkers (alcohol-naive individuals or current abstainers) or individuals with no experience drinking 5 or more drinks on one occasion in their lifetime. Justification: It would be unethical to administer alcohol to individuals that do not drink alcohol. [Based on: medical history].
7. Current or prior history of alcohol-induced flushing reactions, including rapid reddening of the face, rapid heart rate and breathing, and nausea after 1 or 2 drinks. Justification: It would not be safe to administer alcohol to individuals with the highly aversive flushing response to alcohol. [Based on: alcohol flushing questionnaire].
8. Positive result on urine drug screen or positive breathalyzer during screening visit. Positive urine drug screen or breathalyzer reading during more than 1 study visit will result in participant withdrawal from the study. Justification: Current or recent exposure to alcohol or drugs of abuse could impact brain function and alcohol response. [Based on: laboratory tests and breathalyzer test].
9. History of significant withdrawal symptoms or presence of clinically significant withdrawal symptoms (Clinical Institute Withdrawal Assessment (CIWA) score > 8) at screening. Justification: Withdrawal symptoms would be indicative of alcohol use disorder, which is already an exclusion criterion. Additionally, withdrawal symptoms would be a major safety concern for participants, and a major confound in the assessment of alcohol response and brain function. [Based on: CIWA assessment].
10. Medication exclusion criteria: [Based on Medical history and physical exam, Additional History Form].

    * Use of prescription or OTC medication known to interact with alcohol 2 weeks prior to screening or screening update visit. These include but may not be limited to: isosorbide; nitroglycerine; benzodiazepines; warfarin; anti-depressants such as amitriptyline, clomipramine and nefazodone; anti diabetes medications such as glyburide, metformin and tolbutamide; H2-antagonists for heartburn such as famotidine, cimetidine and ranitidine; muscle relaxants; anti-epileptics including phenytoin and phenobarbital; codeine and opioid analgesics including Darvocet, Percocet and hydrocodone.
    * Regular (more than once a week) or prescribed use of antihistamines, pain medicines, and anti-inflammatories such as aspirin, ibuprofen, acetaminophen, celecoxib, and naproxen, and unable to refrain from these medications for 48 hours prior to study visits.NOTE: Seasonal use of antihistamines is not-exclusionary unless participants are unable to refrain from these medications for

      48 hours prior to study visits.
    * Use of medications known to inhibit or induce enzymes that metabolize alcohol for 4 weeks prior to screening or screening update visit. These include chlorzoxazone, isoniazid, metronidazole, and disulfiram.
    * Use of drugs known to affect hemodynamic response 2 weeks prior to screening or screening update visit. These include antihypertensives, insulin, and thyroid medications.
11. Exclusion criteria for MRI:

    * Left-handedness (Edinburgh Handedness Scale). Justification: To avoid lateralized effects on brain function measures and reduce potential variance in MRI signals.
    * Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head (including but not limited to pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments).
    * Fear of enclosed spaces. Justification: To minimize risk and discomfort.
    * Inability to lie comfortable on back for up to 2 hours in the MRI scanner. Justification: To minimize risk and discomfort.

    [Based on: MRI Safety Screening Questionnaire, Additional History Form]
12. Exclusion criteria for persons of childbearing potential:

Justification: To minimize the risk of administering alcohol to pregnant or nursing persons, given the known effects of alcohol exposure on fetuses and infants.

* Pregnant [Based on: urine beta-hCG test at screening]. Persons of childbearing potential must also test negative on urine beta-hCG test at the start of every study visit.
* Breast-feeding [Based on: Medical history and physical exam].

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoints: IV alcohol self-administration measures Peak breath alcohol concentration (BrAC), number of alcohol infusions received. | 2 YEARS
  The Peak BrAC and number of infusions are direct measures of alcohol exposure and amount consumed during the laboratory session.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay A Ramchandani, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002228-AA.html